CLINICAL TRIAL: NCT04053231
Title: Hepatocarcinoma Recurrence on the Liver Study - Part2
Acronym: HERCOLES2
Status: Not yet recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Fabrizio Romano, Professor of Surgery, University of Milano Bicocca
Other Study IDs: HERCOLES-2
Record Dates: First submitted 2019-07-06; First posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Liver Cancer; Surgery; Recurrence Tumor; Cirrhosis
Keywords: liver; hcc; hepatocarcinoma; surgery; redo surgery; recurrence; cirrhosis
MeSH Terms: conditions — Liver Neoplasms; Recurrence; Fibrosis; Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: liver resection — all type of liver surgical procedures

SUMMARY:
Rationale for the trial. To evaluate the impact of surgery on hepatocarcinoma recurrence. Thus, to evaluate the impact of different clinical, radiological, histopathological variables on recurrence after surgical treatment. The nature of this study will allow to observe, over time, the distribution of the considered collection variables, allowing a strictly observational monitoring of possible associations able to suggest models or interpretations, which can then be the basis for the construction of prospective and randomized studies.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is 1 of the 5 most common malignancies worldwide and the third most common cause of cancer related mortality of 500,000 deaths globally every year. Although more common in East Asia, the incidence of HCC is increasing in the Western world. Hepatic resection is the first-line therapeutic option and it is accepted as a safe treatment with a proven impact on prognosis, with a low operative mortality as the result of advances in surgical techniques and perioperative management. Nevertheless, surgical resection is applicable in only about 20% to 30% of patients with HCC, since most have poor hepatic reserve function caused by underlying chronic liver disease and multifocal hepatic distributions of HCC.

Although hepatic resection is one of the curative treatments for hepatocellular carcinoma, the recurrence rate of HCC even after curative resection is quite high, estimated to be approximately 50 % during the first 3 years and more than 70 % during the first 5 years after curative resection, and so the postoperative long term results remain unsatisfactory. In this scenario the role of liver transplantation has been, in the last years, predominant, due to the ability of transplant to reduce disease recurrence, because of the treatment of liver cirrhosis associate to HCC which represent the most important driver to recurrence. Otherwise the scarcity of organ source has been a boost to the spread of liver resection, not only confined in the boundary taken into account in the BCLC algorithm (guidelines endorsed by EASL and AASLD), but even in patients considered not suitable for curative treatment as well as liver resection.

Although surgical treatment has been adopted in the last years in more patients outside the Guidelines with satisfactory results in term of mortality, morbidity and Short term oncological outcomes, the limits of this approach remain the long term disease free survival.

Risk factor for recurrence has been yet identified in the last years as hcc dimension, grading, microvascular invasion and satellitosis. The evidence that these two prognostic factors could negatively impact on the long term prognosis enhancing the risk of recurrence, has led many Author to propose anatomical resection (segmental resection) as the ideal surgical treatment to reduce these risks in HCC patients. Otherwise literature results are in conflict regarding the real benefit of this approach. In fact in many patients with HCC and underlying cirrhosis the anatomical approach is not feasible due to the risk of postoperative liver failure. So a parenchyma-sparing technique has been developed and compared to anatomical resection in term of oncological outcomes. Even if radiological and clinical pictures seems to predict the prognosis of resected HCC, the pathophysiology behind the recurrence is still unclear.Currently, data suggests two type of recurrence presentation: intrahepatic metastasization (IM) and multicentric occurrence (MO) of de novo HCC based on the precancerous status of the remnant diseased liver. Several effort has been done to preoperatively identified the 2 pattern of recurrences. Genetical studied has been performed, especially in eastern countries to better clarify and understand the impact of the 2 phenomena. In the japanese guidelines are described histo-pathological hallmarks able, in retrospect, to define the type of recurrence, metastases or de novo tumor. Moreover, several recent studies including a metanalysis, seems to show that de novo recurrence could have a better prognosis when approached surgically, with a significant improvement in overall and disease-free survival rates. The model of HCC recurrence is not yet well clarified as well as the best treatment of hcc recurrence. On these data is based the proposal to create an Italian study project on surgical treatment and surgical outcomes of hepatocellular carcinoma in term of disease free survival. The idea growth up from the finding that, although the curative intent of surgical approach, results are not so satisfactory and it seems to not ameliorate the long term patient's prognosis and long term disease-free outcome without the need for therapies, conditioning the real everyday life of patient. In Italy is not yet present a study group that draw together the experience of surgical centers with low,medium or high volume of surgical procedures on HCC, with the intent to offer radical cure through surgery as the first choice treatment. The intent is to collect Big Data through a common database, with high power of analysis and high scientific impact, to better understand the mechanism which regulate HCC recurrence and to identify the best clinical treatment option for these patients.

ELIGIBILITY:
Inclusion Criteria:

* No age limit.
* Hepatocarcinoma diagnosis confirmed at histological specimen
* Every single patients with first HCC diagnosis or with a recurrence/persistence disease evaluated and treated with surgery at the participating center.
* the assessment for patient enrollment must have been performed starting from 02/02/2019.

Exclusion Criteria:

* Surgery as a downstaging therapy for transplant
* Patients treated with surgery in case of not-curative intent (palliation, best supportive care, etc).
* Histopathological specimen of combined liver primary neoplasms (e.g. "hepatocholangiocarcinoma'').
* Patients with other tumors in the previous past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated by surgery for HCC
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2034-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free-Survival | 15 years of follow-up
  Disease Free Survival: the time between surgery and event of recurrence or death measured in months. If no event, patients will be censored at the last available follow-up date.
Overall Survival | 15 years of follow-up
  The time from surgery to death measured in months. If no event, patients will be censored at the last available follow-up.

SECONDARY OUTCOMES:
Localization of the recurrence | 15 years of follow-up
  Presence of relapse disease on the surgical cut surface rather than at distance
Number of redo-surgery | 15 years
  Number of patients who experienced a recurrence after first surgery and has been submitted to a redo-surgery procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Romano, MD, Principal Investigator — University of Milan-Bicocca; Simone Famularo, MD, Principal Investigator — University of Milan Bicocca
Locations (19):
- Italy (19):
  - Chirurgia Rubino - Policlinico di Bari, Bari
  - Ospedale Maggiore- AUSL, Bologna
  - Chirurgia Generale Bolzano, Bolzano
  - Fondazione Poliambulanza - Istituto Ospedaliero, Brescia
  - Spedali Civili, Brescia
  - Chirurgia Generale Ospedale Pierantoni - Morgagni, Forlì
  - Ospedale A. Manzoni - ASST Lecco, Lecco
  - ASST-Mantova, Mantova
  - Asst-Fbf-Sacco Polo Universitario H. Sacco Chirurgia 2, Milan
  - IRCCS Osp. San Raffaele, Divisione Chirurgia Generale Epatobiliare, Milan
  - Policlinico di Monza, Monza
  - UOS Chirurgia Oncologica ad inidirzzo epato-bilio-pancreatico, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario A. Gemelli, IRCCS, Rome
  - Irccs Istituto Nazionale Tumori Regina Elena, Rome
  - Humanitas Research Hospital, Rozzano
  - Ospedale San Paolo, Savona
  - Chirurgia 4 Ospedale Ca'Foncello, Treviso
  - Chirurgia Epatobiliare Università degli studi di Verona, Verona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: All the informations and protocol are available at the website — http://www.hercolesgroup.eu